CLINICAL TRIAL: NCT03284619
Title: First-In Man (FIM) Study MR-Linac
Acronym: FIM MR-Linac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nucletron Operations BV (Industry)
Collaborators: Factory CRO for Medical Devices B.V. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MR-Linac-CIP-001 Version 2.0; NL60984.041.17 (Other: CCMO)
Record Dates: First submitted 2017-06-22; First posted 2017-09-15 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Bone Metastases

STUDY DESIGN:
Intervention Model Description: Proof of concept including accuracy and safety aspects according to R-IDEAL stage 1 criteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): Single arm study, 5 patient with bone metastasis will be enrolled for palliative treatment with the Magnetic resonance imager linear accelerator (MR-Linac).
  Interventions: Device: Magnetic resonance imager linear accelerator

INTERVENTIONS:
Device: Magnetic resonance imager linear accelerator — The MR linear accelerator (MRL) integrates a radiotherapy accelerator and a diagnostic quality 1.5T MRI, enabling soft-tissue visualization during the actual radiation delivery for improved targeting. This enables on-line treatment optimization for precise radiation delivery. Better visualization of the tumour targets and the surrounding healthy tissues, at the exact moment of treatment, makes it possible to adapt the dose to the actual anatomy while optimally sparing normal tissues.
  Other Names: MR-Linac; Unity

SUMMARY:
Investigational device is the Magnetic resonance imager linear accelerator. Five (5) patients with bone metastases will be treated with palliative intention in this study. The goal is to confirm the pre-clinically demonstrated technical accuracy and safety of the newly developed MR-Linac in the clinical setting.

DETAILED DESCRIPTION:
This is a single center prospective proof of concept study including accuracy and safety aspects according to R-IDEAL stage 1 criteria. Five (5) patients with bone metastases will be treated with palliative intention in this study. Treatment will consist of a single fraction.

The MR linear accelerator (MRL) integrates a radiotherapy accelerator and a diagnostic quality 1.5T MRI, enabling soft-tissue visualization during the actual radiation delivery for improved targeting. This enables on-line treatment optimization for precise radiation delivery. Better visualization of the tumour targets and the surrounding healthy tissues, at the exact moment of treatment, makes it possible to adapt the dose to the actual anatomy while optimally sparing normal tissues.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a patient must meet all of the following criteria:

* Painful bone metastases in the lumbar spine
* Radiographic evidence of bone metastases
* Histologic proof of malignancy (primary carcinoma)
* Karnofsky Performance Score ≥ 50
* Age ≥ 18 years
* Able to provide written informed consent

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Prior radiation therapy within the region planned to be irradiated
* Contraindication for MRI according to screening protocol radiology department UMCU (e.g. cardiac pacemakers, and defibrillators, artificial heart valves or cochlear implants, https://richtlijn.mijnumc.nl/Beeld/MRI/Paginas/MRI-Veiligheid-Contra-indicaties.aspx
* Claustrophobia
* Standard systemic anti-cancer therapy or radionuclide therapy within 48 hours before or after treatment.
* Any other type of not standard systemic anti-cancer treatment, except for endocrine treatment.
* Unstable spine requiring surgical stabilization
* Neurological deficit due to bone metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Safety of the treatment system (a dose distribution accuracy ≤ 5% will be considered acceptable). Incidence of acute toxicity (CTCAE grade 2 are higher) and incidence of Serious (unexpected) Adverse Events will be measured. | During treatment (Day 0). For patient safety patients will be contacted at day 1, week 2 and week 12 after treatment.
  Safety of the system: System behaves in accordance with the workflow and risk mitigation plan, Dosimetric safety: An independent dosimetry check before start irradiation (Oncentra) and an independent dosimetry during irradiation (second chamber) will be used. For the overall process a dose distribution accuracy ≤ 5% will be considered acceptable.
  Patients safety: by reporting any acute toxicity > grade 2 (according CTCAE version 4.0 for acute toxicity) and any Serious (Unexpected) Adverse Events (S(U)AE) within 12 weeks after treatment
Geometrical accuracy of targeting by online MR imaging | During treatment (day 0)
  Geometrical accuracy: will be checked online by using the MRI in combination with VolumeTool visualization and off-line by comparison of the EPID beam data with the prescribed beam data. A positioning error of ≤ 5 mm will be considered acceptable

SECONDARY OUTCOMES:
Descriptive analysis of the clinical workflow by keeping a log book for the entire procedure. | During treatment (day 0)
  Feasibility of the clinical workflow: by keeping a log book for the entire procedure. The validation of radiation delivery includes assessing the hardware performance and the See-Plan-Treat work flow for on-line MRI guided adaptive radiotherapy.
Patients comfort | immediately after treatment (day 0)
  Patient comfort during the MR-Linac treatment: by patient questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ina Jürgenliemk-Schulz, MD, PhD, Principal Investigator — UMCU
Locations (1):
- University Medical Centre Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No